CLINICAL TRIAL: NCT06102707
Title: The Efficacy and Safety of Fluzopril Combined With Apatinib in Maintenance Treatment of Platinum Resistant Recurrent Ovarian Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202210-045
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzopril Combined With Apatinib Group (Experimental)
  Interventions: Drug: Fluzopril Combined With Apatinib

INTERVENTIONS:
Drug: Fluzopril Combined With Apatinib — Fluzopril Capsules 100mg po bid Apatinib Mesylate Tablets 250mg po qd

SUMMARY:
Ovarian cancer is the most lethal gynecological malignancy, posing a serious threat to women's health worldwide.Platinum resistant ovarian cancer is the biggest challenge faced by gynecological oncologists.Exploring more effective treatment options and how to delay the recurrence of platinum resistant recurrent ovarian cancer remains a challenging issue in clinical treatment.The main goal of this trial is to evaluate the effectiveness and safety of fluzopril combined with apatinib in maintenance treatment of platinum resistant recurrent ovarian cancer patients by evaluating progression free survival (PFS).Fifty patients with advanced ovarian cancer who underwent platinum resistant recurrent chemotherapy and assessed no disease progression were enrolled in the study, and maintenance treatment was performed with fluzopril combined with apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.
2. Female, age ≥ 18 years old (calculated based on the date of signing informed consent).
3. High grade (or medium to low differentiation) serous ovarian cancer, fallopian tube cancer, or primary peritoneal cancer confirmed by pathology; Or moderately or poorly differentiated ovarian endometrioid adenocarcinoma. Disease progression occurred within 6 months (182 days) of the last platinum containing chemotherapy.
4. Received at least 3 cycles of chemotherapy.
5. After the completion of chemotherapy treatment, it is evaluated as non disease progression and must be randomly enrolled within 6 weeks after the last dose of chemotherapy is administered.
6. Must be able to provide tumor tissue samples fixed with formalin and embedded in paraffin (FFPE).
7. The Eastern Cooperative Oncology Group score is 0-1.
8. The function of important organs meets the following requirements (no blood components or cell growth factors are allowed to be used within the first 14 days of randomization):absolute neutrophil count ≥ 1.5 × 109/L; Platelets ≥ 100 × 109/L; Hemoglobin ≥ 90g/L;Serum albumin ≥ 3g/dL;Bilirubin ≤ 1.5 times ULN;ALT and AST ≤ 3 times ULN; Serum creatinine ≤ 1.5 times ULN.
9. Patients with potential fertility need to use at least one medically approved contraceptive method (such as an intrauterine device or condom) during the study treatment period and within 3 months after the end of the study treatment period, and must have a negative serum HCG test within 72 hours before randomization; And it must be non lactating.

Exclusion Criteria:

1. Subjects had other malignant tumors in the past (within 5 years) or at the same time, except for cured skin basal cell carcinoma, cervical carcinoma in situ and breast cancer that had no recurrence for more than 3 years after the completion of radical surgery.
2. Previously used both PARP inhibitors and small molecule VEGF inhibitors, including but not limited to olaparib, nilaparib, arotinib, apatinib, etc; Single drug treatment can be included in the group.
3. Patients with untreated central nervous system metastasis who have previously received systemic or curative brain or meningeal metastasis treatment (radiotherapy or surgery), and have been confirmed stable by imaging for at least 1 month, and have stopped systemic hormone therapy (dosage>10mg/day of prednisone or other effective hormones) for more than 2 weeks, without clinical evidence, can be included.
4. Patients who have recently experienced intestinal obstruction or gastrointestinal perforation (within 3 months).
5. Patients who are unable to swallow tablets normally or have gastrointestinal dysfunction, as determined by the researchers, may affect drug absorption.
6. Patients with clinical symptoms of cancerous ascites or pleural effusion who require puncture or drainage, or who have received ascites or pleural effusion drainage within the first 3 months of randomization.
7. Patients with clinically uncontrolled cardiac symptoms or diseases, such as NYHA grade 2 or above heart failure, unstable angina pectoris, myocardial infarction within 1 year, clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention, and QTc>470ms.
8. Patients with hypertension who cannot achieve good control after treatment with antihypertensive drugs (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg).
9. Any bleeding event with a severity rating of 2 or above in CTCAE 5.0 within the first 4 weeks of randomization.
10. Previous or current history of idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, tissue pneumonia (such as bronchitis, occlusive vasculitis), drug-induced pneumonia, or screening stage CT showing active pneumonia.
11. Individuals with abnormal coagulation function (INR>1.5 or prothrombin time>ULN+4 seconds), bleeding tendencies, or undergoing thrombolytic or anticoagulant treatment are allowed to receive low-dose low-molecular-weight heparin or oral aspirin for prophylactic anticoagulant treatment during the trial period.
12. There have been incidents of arterial/venous thrombosis within the first 6 months of randomization, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep venous thrombosis, and pulmonary embolism.
13. Patients with a history of hereditary or acquired hemorrhagic disease or coagulation disorders. Within the first 3 months of randomization, there were significant clinically significant bleeding symptoms or clear bleeding tendencies, such as gastrointestinal bleeding, hemorrhagic gastric ulcers, etc.
14. Subject has active infection or unexplained onset of ≥ 38.5 ° C within 7 days prior to randomization.
15. Subjects have congenital or acquired immune deficiency (such as HIV infected persons), or active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA ≥ 500IU/ml; hepatitis C reference: HCV antibody positive and HCV copy number>upper limit of normal value).
16. Patients who have received surgery, radiation therapy, chemotherapy, and endocrine therapy before randomization for less than 4 weeks after treatment completion; Adverse events caused by previous treatment (excluding hair loss) that have not recovered to ≤ 1 level (CTCAE 5.0).
17. Patientss who may receive other systemic anti-tumor treatments or plan to undergo ovarian cancer reduction surgery during the study period.
18. According to the judgment of the researchers, there are other factors that may lead to the forced termination of this study, such as other serious illnesses (including mental illness) requiring concurrent treatment, serious laboratory test abnormalities, accompanied by family or social factors, which may affect the safety of the subjects, or the collection of data and samples.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease progression free survival | 36 months
  Disease progression free survival (PFS) evaluated by researchers based on RECIST 1.1 criteria